CLINICAL TRIAL: NCT06493474
Title: Effect of Peer Assisted Breastfeeding Education Program (PABEP) on Breastfeeding Self-Efficacy and Breastfeeding Levels: Randomized Controlled Study
Brief Title: Peer Assisted Breastfeeding Education Program
Acronym: PABEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tasdemir, Assistant Professor, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAKU24-01
Record Dates: First submitted 2024-06-26; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PABEP group (Experimental): In the research, first of all, breastfeeding training will be given to a nurse mother who has given birth. After this training, the nurse will convey to the mothers the problems she has experienced and coping methods at the end of each training period during the training that the researcher will give to the mothers.
  Interventions: Other: Education
- Control Group (Active Comparator): They will only receive the routine training provided by the application center.
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Education — PEER ASSISTED BREASTFEEDING EDUCATION PROGRAM
  Arms: PABEP group
Other: Routine Care — Non education program only routine care
  Arms: Control Group

SUMMARY:
It was aimed to evaluate the effect of the Peer Supported Breastfeeding Education Program given during the antenatal period on the breastfeeding knowledge and attitude levels, breastfeeding self-efficacy and breastfeeding levels of postpartum women. For this purpose, the hypotheses created in our study are as follows.

1. H1: Breastfeeding knowledge and attitudes of mothers in the PABEP group are significantly higher than those in the control group.
2. H1: Breastfeeding proficiency levels of mothers in the PABEP group are significantly higher than those in the control group.
3. H1: Breastfeeding success of mothers in the PABEP group is significantly higher than the control group, according to the breastfeeding evaluation results.

ELIGIBILITY:
Inclusion Criteria:

* being in the antenatal period
* having their first pregnancy
* not having received breastfeeding counseling before.

Exclusion Criteria:

* mothers with previous birth history
* previously educated women

Max Age: 36 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — women aged 20-45 in the antenatal period
Enrollment: 170 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy | Research data will be collected during training before birth and at 1 and 4 weeks after birth.
  It is a scale consisting of 33 items developed by Dennis (1999). The scale prepared as a five-point Likert type; (1) I never trust myself, (2) I don't trust myself very much, (3) I sometimes trust myself, (4) I trust myself most of the time, (5) I always trust myself. As the total score on the scale increases, breastfeeding self-efficacy also increases. The lowest score is 33 and the highest score is 165.

SECONDARY OUTCOMES:
breastfeeding success | Research data will be collected during training before birth and at 1 and 4 weeks after birth.
  The scale consists of six questions and scoring is based on mothers' answers to the questions. The first question is about the baby's starting state of feeding (deep sleep, sleepy, calm-awake, crying). This question is not included in the scoring. The next four questions are about searching and the baby's sucking behavior. Each question is evaluated between 0-3 points and the highest score is 12. The score range in effectively fed babies is 10-12 points. Babies who breastfeed quite successfully when encouraged are given 7-9 points and are considered moderately effective. Babies who do not start feeding upon warning, do not seek nutrition, or breastfeed for short periods are given a score of 0-6. In the last question, mothers record their feelings during feeding (very satisfied, satisfied, not very satisfied, not satisfied). This question is not included in the scoring and is evaluated separately.

CONTACTS AND LOCATIONS:
Overall Officials: Halil HI Taşdemir, PhD, Study Director — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
data contains confidentiality